CLINICAL TRIAL: NCT07276282
Title: Effects of Ziltivekimab Versus Placebo on Coronary Atherosclerosis in Patients With Acute Myocardial Infarction. A Serial, Multivessel, Intravascular Ultrasound, Near-infrared Spectroscopy and Optical Coherence Tomography Imaging Study
Brief Title: Effects of Ziltivekimab on Coronary Atherosclerotic Burden in Patients With Acute Myocardial Infarction
Acronym: ZEPHYR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ECRI bv (Industry)
Collaborators: Novo Nordisk A/S (Industry); Insel Gruppe AG, University Hospital Bern (Other); Cardialysis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECRI-16; 2024-520364-34-00 (EU CTIS Number); NN6018-8195 (Other: Novo Nordisk A/S)
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Acute Myocardial Infarction (AMI); Coronary Atherosclerosis of Native Coronary Artery
Keywords: IL-6 inhibition; atherosclerosis; acute myocardial infarction; anti-inflammatory; intracoronary imaging
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — ziltivekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clinical Research Organization, Data Coordinating Center, Core Laboratories
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ziltivekimab Arm (Experimental): Participants will receive Ziltivekimab subcutaneously once per month
  Interventions: Drug: Ziltivekimab
- Placebo Arm (Placebo Comparator): Participants will receive placebo subcutaneously once per month
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ziltivekimab — Ziltivekimab is administered subcutaneously (i.e., under the skin) once per month added to standard of care.
  Arms: Ziltivekimab Arm
Drug: Placebo — Placebo is administered subcutaneously (i.e., under the skin) once per month added to standard of care.
  Arms: Placebo Arm

SUMMARY:
Despite improvements in the treatment, coronary artery disease (CAD) remains one of the leading causes of death worldwide. Around 20% of people who have suffered a heart attack (myocardial infarction) need to be hospitalized again within a year, and 10% experience another heart attack. Despite currently available medication, patients remain at risk of further episodes after a heart attack. Scientists have discovered that inflammation in the body plays a decisive role in the development and narrowing of arterial blockages (atherosclerosis). This study aims to investigate whether a new treatment that reduces inflammation can help improve the arteries of patients with CAD.

This study will examine whether blocking certain inflammation-related substances with a new medicinal product called ziltivekimab affects the buildup and composition of plaques (fatty deposits) in the coronary arteries. Special imaging diagnostic techniques will be used to look inside the arteries and check whether the treatment helps reduce the narrowing caused by dangerous plaques, which can lead to future heart attacks.

This is a clinical study in which participants are randomly divided into two groups (randomization): one group will receive the new treatment ziltivekimab and other group will receive a placebo (a harmless substance with no active ingredients). Both groups will continue to receive standard treatment for heart attacks. The study lasts approximately 15 months per participant.

The full scientific title of the trial is: Effects of ziltivekimab versus placebo on coronary atherosclerosis in patients with acute myocardial infarction. A study with serial multi-vessel imaging obtained using intravascular ultrasound, near-infrared spectroscopy, and optical coherence tomography techniques.

DETAILED DESCRIPTION:
Despite advances in cardiovascular care and preventive treatments, coronary artery disease (CAD) still represents the leading causes of death worldwide. Almost one fifth of patients with acute myocardial infarction (MI) suffer from rehospitalization within 1 year and 10% from recurrent MI. This residual cardiovascular risk persists regardless of optimal medical therapy with contemporary pharmacologic treatments including lipid lowering drugs, suggesting that this excess risk is mediated through pathways not yet directly addressed by current management. Inflammation is now a well-acknowledged major contributor to atherosclerosis development and plaque progression/instability, with both the innate (monocyte-derived macrophages) and the acquired immune system (T-cells) thought to be involved. Within atherosclerotic human plaques, activated monocyte-derived macrophages, specialized CD4+ and CD8+ T-cells produce a wide array of chemokines and cytokines with pro-inflammatory effects.

Despite a growing body of evidence that has confirmed anti-inflammatory therapy as a new cornerstone opportunity to reduce effectively the residual cardiovascular risk in CAD patients with CAD treated with optimal medical therapy, the direct effect of these therapies on atherosclerosis extension and composition is largely unknown. Convincing experimental evidence has raised the translational hypothesis of a direct favourable effect of IL-6 inhibition on plaque biology and stabilization. However, in-human data regarding the mechanistic role of anti-IL-6 agents on coronary atherosclerosis are lacking so far.

The purpose of this study is to investigate for the first time the in-vivo effects of IL-1/IL-6 pathway inhibition on coronary plaque morphology and composition in patients with CAD. Serial multi-vessel images obtained with multimodality intracoronary imaging will allow for a comprehensive evaluation of presumed high risk atherosclerotic features such as plaque burden, fibrous cap thickness, lipid content and local inflammation. An intracoronary serial imaging study may elucidate the exact pathophysiological underpinnings of atheroprotection beyond lipid lowering therapy and assess whether an effective anti-inflammatory therapy can improve the atherosclerotic profile of patients with CAD.

This is an interventional, randomised, parallel-group, double-blind, placebo-controlled, multi-centre, multi-national study designed to evaluate the effects of ziltivekimab versus placebo (randomised 1:1), both administered s.c. once-monthly and added to standard of care, on change in percent atheroma volume (PAV) as well as change in maxLCBI and fibrous cap thickness. The initial dose of ziltivekimab s.c./placebo to be administered at randomisation which is as early as possible and latest within 48 hours after the index PCI procedure, followed by once-monthly administration during the treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

* Informed consent obtained before any study-related activities.
* Age 18 years or above at the time of providing informed consent.
* Acute myocardial infarction, with at least one coronary segment (culprit lesion) treated with PCI.
* At least two major native coronary arteries each meeting angiographic criteria for intracoronary imaging immediately following the qualifying PCI procedure.

Key Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Known allergy to contrast medium, heparin, aspirin, ticagrelor or prasugrel.
* Female of childbearing potential.
* Left-main disease.
* Three-vessel disease.
* History of coronary artery bypass surgery.
* TIMI flow <2 of the infarct-related artery after PCI.
* Unstable clinical status (hemodynamic or electrical instability.
* Significant coronary calcification or tortuosity deemed to preclude IVUS, NIRS and OCT evaluation.
* Uncontrolled cardiac arrhythmia.
* Severe kidney impairment.
* Active liver disease or hepatic dysfunction.
* Current use of anti-IL-6 products or anticipated use of such drugs any time during the study.
* Use of systemic immunosuppressive drugs or disease modifying anti-rheumatic drugs or anticipated chronic use of such drugs any time during the study.
* Known, or suspicion of, active infection or major hematologic, metabolic, or endocrine dysfunction in the judgment of the Investigator
* History of recurrent serious infections.
* Use of preventive systemic antibiotics, systemic antivirals, or systemic antifungals.
* Known (acute or chronic) hepatitis B or hepatitis C
* Planned surgery within 12 months from the time of screening.
* History of cancer within the past 5 years, except for adequately treated basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, low risk prostate cancer, or carcinoma in situ/high grade prostatic intraepithelial neoplasia (PIN) at the discretion of the investigator.
* Estimated life expectancy less than 2 years
* Received a live or attenuated-live vaccine product within 4 weeks of study intervention administration or expected to receive a live or attenuated-live vaccine product during the treatment period.
* Major cardiac surgical within the past 60 days or any major surgical procedure planned at the time of randomisation or as treatment for the current AMI (CABG).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in percent atheroma volume | From randomization (week 0) to end-of-study (52-week)
  Change in percent atheroma volume (PAV) as determined by greyscale intravascular ultrasound (IVUS) in matched regions of interest. Theoretical change is between -100% to +100%. Typical range around -2% to +2%. A lower (more negative) change in PAV is better.

SECONDARY OUTCOMES:
Maximum lipid core burden index | From randomisation (week 0) to end-of-study (52-week)
  Change in maximum lipid core burden index (LCBI) in any 4-mm segment (maxLCBI4mm) as determined by NIRS in matched regions of interest. Theoretical range is between -1000 to +1000. Typical range around -250 to +250. A lower (more negative) change is better.
Minimal fibrous cap thickness | From randomisation (week 0) to end-of-study (52-week)
  Change in minimal fibrous cap thickness as determined by optical coherence tomography (OCT) in matched regions of interest. Theoretical range is between -500 µm to +500 µm. Typical range around -50 µm to +110 µm. A higher (positive) change is better; it indicates fibrous cap thickening (increased plaque stability).

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Räber, MD, PhD, Principal Investigator — Cardiology Department, Bern University Hospital, Inselspital Bern, Switzerland; Ernest Spitzer, MD, Study Director — European Cardiovascular Research Institute
Locations (1):
- Bern University Hospital, Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No